CLINICAL TRIAL: NCT02799706
Title: Phase IIIb Randomized Trial Comparing Irradiation Plus Long Term Adjuvant Androgen Deprivation With GnRH Antagonist Versus GnRH Agonist Plus Flare Protection in Patients With Very High Risk Localized or Locally Advanced Prostate Cancer. A Joint Study of the EORTC ROG and GUCG
Brief Title: Trial Comparing Irradiation Plus Long Term Adjuvant Androgen Deprivation With GnRH Antagonist Versus GnRH Agonist Plus Flare Protection in Patients With Very High Risk Localized or Locally Advanced Prostate Cancer
Acronym: PEGASUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1414
Record Dates: First submitted 2016-05-17; First posted 2016-06-15 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; GnRH antagonist; GnRH agonist; radiation therapy; very high risk localized prostate cancer; locally advanced prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GnRH agonist + radiation therapy (RT) (Active Comparator): As the study investigates the effect of a drug given concomitantly to radiotherapy, all patients will be treated with the same treatment technique and target dose. The preferred treatment technique is intensity modulated radiotherapy (IMRT) + A GnRH-agonist will be given for the duration selected for each patient.
  A non-steroidal anti-androgen (e. g. flutamide, bicalutamide) will be given orally one week before the first injection of the GnRH agonist and will be continued for no longer than 8 weeks to protect against flare.
  Dose may vary due to availability of different brand names and pharmaceutical forms The start of antiandrogen must be registered as day 1 of treatment in the GnRH agonist arm.
  Interventions: Drug: approved GnRH agonist; Radiation: Radiotherapy
- GnRH antagonist + radiation therapy (RT) (Experimental): As the study investigates the effect of two drugs given concomitantly to radiotherapy, all patients will be treated with the same treatment technique and target dose. The preferred treatment technique is intensity modulated radiotherapy (IMRT) +a GnRH antagonist will be given for a predefined duration of 18, 24, or 36 months as per institution policy.
  Each institution has to adhere to the chosen duration of treatment for all patients throughout the study
  Interventions: Drug: Degarelix; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Degarelix — a GnRH antagonist will be given for a predefined duration of 18, 24, or 36 months as per institution policy
  Arms: GnRH antagonist + radiation therapy (RT)
Drug: approved GnRH agonist — A non-steroidal anti-androgen (e. g. flutamide, bicalutamide) will be given orally one week before the first injection of the GnRH agonist and will be continued for no longer than 8 weeks to protect against flare.Dose may vary due to availability of different brand names and pharmaceutical forms The start of antiandrogen must be registered as day 1 of treatment in the GnRH agonist arm.
  Arms: GnRH agonist + radiation therapy (RT)
Radiation: Radiotherapy — .As the study investigates the effect of two drugs given concomitantly to radiotherapy, all patients will be treated with the same treatment technique and target dose. The preferred treatment technique is intensity modulated radiotherapy (IMRT)

SUMMARY:
The primary objective of the trial is to assess if GnRH antagonists in combination with external beam radiation therapy improve progression free survival (progression that can be biological, clinical, or death) compared to GnRH agonists in combination with external beam radiation therapy.

Secondary objectives include:

* documentation of effect of GnRH antagonists on clinically significant cardiovascular events in the subgroup of patients at high risk of such events at baseline;
* documentation of side effects and quality of life, I-PSS and urinary tract infections;
* assessment of relative treatment effect on secondary efficacy endpoints (clinical progression, time to next line of systemic therapy, time on therapy, overall and cancer specific survival) and on PSA at 6 months after end of RT.

DETAILED DESCRIPTION:
Phase IIIb randomized stratified open-label comparative 2-arm superiority study with a pre-set non-inferiority boundary.

Registered GnRH antagonists, degarelix, will be given at the dose of 240 mg given as two subcutaneous injections of 120 mg at a concentration of 40 mg/mL on day 1, followed by 80 mg given as one subcutaneous injection at a concentration of 20 mg/mL every 28 days (±2 days).

External beam radiotherapy (EBRT) to a total dose of 78-80 Gy, delivered as one daily fraction, five days a week, started between d1 and months 6 of the androgen deprivation therapy as per institution policy. The irradiation is the same as in the reference therapy arm.

The minimum duration of androgen deprivation with GnRH agonist or antagonist therapy is 18 months.

For each patient, the duration of therapy must be elected upfront by the treating physician among three possible options: 18, 24 or 36 months. The institution shall also declare upfront the duration of the neoadjuvant treatment they intend to deliver to each patient (between 0 and 6 months).

The primary endpoint is progression-free survival defined as the time in days from randomization to death, clinical or biochemical progression, whichever comes first.

Where

* PSA progression based on Phoenix definition, i.e. a rise by 2 ng/mL or more above the nadir PSA (Ref. 17) confirmed by a second value measured minimum 3 months later
* Clinical progression is defined as onset of obstructive symptoms requiring local treatment and demonstrated to be caused by cancer progression or evidence of metastases detected by clinical symptoms and confirmed by imaging
* Start of another line of systemic therapy in absence of progression
* Death due to any cause

Secondary endpoints:

* Clinical progression-free survival
* Time to next systemic anticancer therapy (including secondary hormonal manipulation)
* Proportion of patients switching from GnRH antagonists to GnRH agonists and total effective duration of treatment with the originally allocated drug.
* Overall survival
* Cancer specific survival
* PSA at six months after completion of RT Safety will be scored by the CTCAE version 4.0. The major safety endpoints in this study are
* the incidence of clinical cardiovascular events - CCE (i.e. arterial embolic or thrombotic events, hemorrhagic or ischemic cerebrovascular conditions, myocardial infarction, and other ischemic heart disease) in patients who had cardiovascular events before entering the trial and in those without such events.
* Incidence of urinary tract infection

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate adenocarcinoma
* PSA ≥ 10 ng/ml and two of the following 4 criteria:
* PSA ≥ 20 ng/ml,
* Gleason sum ≥ 8,
* cN1 (regional LN with a short axis length >10mm by CT scan or MRI) or pathologically confirmed lymph nodes (pN1),
* cT3-T4 (by MRI or core biopsy) (i.e. If PSA≥ 20 ng/ml then only one of the other 3 risk factors is needed)
* M0 by standard imaging work-up (see chapter 6.1.1.1)
* Testosterone ≥ 200 ng/dl
* Adequate renal function: calculated creatinine clearance ≥ 50 mL/min (Appendix D) Magnesium and potassium within normal limits of the institution or corrected to within normal limits prior to the first dose of treatment.
* Patients with prolonged QT-intervals due to prescribed Class IA (quinidine, procainamide) or Class III (amiodarone, sotalol) antiarrhythmic medication must be carefully evaluated for GnRH-agonist or GnRH antagonist use, because these drugs may prolong the QT-interval.
* WHO Performance status 0-1
* Age ≥ 18 and ≤ 80 years
* Participants who have partners of childbearing potential must use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 3 months after last dose of study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Previous use of androgen deprivation therapy (ADT), antiandrogens. 5-alpha reductase inhibitors are allowed if interrupted for more than 6 months prior to entering the study
* History of severe untreated asthma, anaphylactic reactions or severe urticaria and/or angioedema.
* Hypersensitivity towards the investigational drug
* The following biological parameters :AST, ALT, total bilirubin, prothrombin time, serum albumin above upper level of normal range No severe hepatic impairment (Child Pugh C)
* History of gastro-intestinal disorders (medical disorder or extensive surgery) that may interfere with the absorption of the protocol treatment.
* History of pituitary or adrenal dysfunction
* Uncontrolled diabetes mellitus
* History of ulcerative colitis, Crohn's Disease, ataxia, telangiectasia, systemic lupus erythematous, or Fanconi anemia.
* Clinically significant heart disease as evidence myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) class III or IV heart disease or cardiac ejection fraction measurement of < 50 % at baseline
* Coronary revascularization (PCI or multivessel CABG), carotid artery or iliofemoral artery revascularization (percutaneous or surgical procedure) within the last 30 days prior to entering the trial
* Certain risk factors for abnormal heart rhythms/QT prolongation: torsade de pointes ventricular arrhythmias (e.g, heart failure, hypokalemia, or a family history of a long QT syndrome), a QT or corrected QT (QTc) interval >450 ms at baseline, or intake of medications that prolong the QT/QTc interval
* Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg); patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment.
* Prior history of malignancies other than prostate adenocarcinoma (except patients with basal cell, squamous cell carcinoma of the skin), or the patient has been free of malignancy for a period of 3 years prior to first dose of study drug(s). Prior history of bladder cancer excludes the patient.
* Prior radical prostatectomy (TURP or suprapubic adenomectomy for benign prostatic hyperplasia is allowed)
* Prior brachytherapy or other radiotherapy that would result in an overlap of radiotherapy fields
* Any contraindication to external beam radiotherapy
* Patients with significantly altered mental status prohibiting the understanding of the study or with psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule or any condition which, in the opinion of the investigator, would preclude participation in this trial

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 885 (Estimated)
Dates: Start 2017-09-25 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | through study completion, an average of 1 year
  The primary endpoint is progression-free survival defined as the time in days from randomization to death, clinical or biochemical progression, whichever comes first.
  Where
  * PSA progression based on Phoenix definition, i.e. a rise by 2 ng/mL or more above the nadir PSA (Ref. 17) confirmed by a second value measured minimum 3 months later
  * Clinical progression is defined as onset of obstructive symptoms requiring local treatment and demonstrated to be caused by cancer progression or evidence of metastases detected by clinical symptoms and confirmed by imaging
  * Start of another line of systemic therapy in absence of progression
  * Death due to any cause

SECONDARY OUTCOMES:
Clinical progression-free survival | through study completion, an average of 1 year
Time to next systemic anticancer therapy (including secondary hormonal manipulation) | through study completion, an average of 1 year
♦ Proportion of patients switching from GnRH antagonists to GnRH agonists | through study completion, an average of 1 year
♦ Overall survival | through study completion, an average of 1 year
Incidence of clinical cardiovascular events | through study completion, an average of 1 year
  ♦ the incidence of clinical cardiovascular events - CCE (i.e. arterial embolic or thrombotic events, hemorrhagic or ischemic cerebrovascular conditions, myocardial infarction, and other ischemic heart disease) in patients who had cardiovascular events before entering the trial and in those without such events.
♦ Incidence of urinary tract infection | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Boehmer, MD, PhD, Principal Investigator — Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin; Pedro Lara, MD, PhD, Principal Investigator — San Roque University Hospital; Thomas Zilli, MD, PhD, Principal Investigator — Hôpitaux universitaires de Genève - HUG - site de Cluse-Roseraie; Martin Spahn, MD, PhD, Principal Investigator — Group Of Private Clinics Hirslanden - Hirslanden Klinik Zurich
Locations (39):
- Belgium (8):
  - Hopitaux Universitaires Bordet-Erasme - Hopitaux Universitaires Bordet- Institut Jules Bordet, Brussels
  - Hopitaux Universitaires Bordet-Erasme - Hopital Universitaire Erasme, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Hopital De Jolimont, Haine-Saint-Paul
  - AZ Groeninge Kortrijk - Campus Kennedylaan, Kortrijk
  - CHU Ucl Namur - Site Sainte-Elisabeth, Namur
  - Gasthuiszusters van Antwerpen - GasthuisZusters Antwerpen - Sint-Augustinus, Wilrijk
- University Hospitals Copenhagen - Rigshospitalet, Copenhagen, Denmark
- France (10):
  - Clinique de l'Europe, Amiens
  - Centre de radiotherapie Marie Curie, Arras
  - Centre D'Onco. & Radioth. De Haute Energie Du Pays Basque, Bayonne
  - Groupe Radiopole Artois - Centre de Radiotherapie Pierre Curie, Beuvry
  - CHU de Grenoble - La Tronche - Hôpital A. Michallon, Grenoble
  - Centre Leon Berard, Lyon
  - Institut de Cancerologie de l'Ouest (ICO) - Centre Rene Gauducheau, Nantes
  - Assistance Publique - Hopitaux de Paris - La Pitie Salpetriere, Paris
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire
  - Clinique Pasteur-Toulouse-Atrium, Toulouse
- Germany (3):
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Otto-Von-Guericke-Universitaet Magdeburg - Universitaetsklinik, Magdeburg
- Italy (2):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - AUSL Romagna - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
- Spain (11):
  - Fundacion Hospital Alcorcon, Alcorcón
  - Institut Catala d'Oncologia - ICO Badalona - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia), Barcelona
  - Clinica IMQ Zorrotzaurre, Bilbao
  - Hospital General Universitario Santa Lucia, Cartagena
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Complejo Hospitalario A, Pamplona
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Consorci Sanitari De Terrassa, Terrassa
  - Complejo Hospitalario Universitario de Vigo -CHUVI - Hospital Alvaro Cunqueiro, Vigo
- Switzerland (3):
  - Oncology Institute of Southern Switzerland (IOSI) - Oncology Institute of Southern Switzerland - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital, Bern
  - Hôpitaux universitaires de Genève - HUG - site de Cluse-Roseraie, Geneva
- Nottingham University Hospitals NHS Trust - City Hospital, Nottingham, United Kingdom

REFERENCES:
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976